CLINICAL TRIAL: NCT03325361
Title: The Role of Transanal Tube Drainage as A Mean of Prevention of Anastomotic Leakage
Brief Title: The Role of Transanal Tube Drainage as A Mean of Prevention of Anastomotic Leakage Anastomotic Leakage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Pierpaolo Sileri, Professor, University of Rome Tor Vergata
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Transanal Tube Drainage
Record Dates: First submitted 2017-10-24; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Rectal Cancer; Rectal Neoplasms; Anastomotic Leak
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TD (Experimental)
  Interventions: Other: Tube drain insertion
- NTD (No Intervention)

INTERVENTIONS:
Other: Tube drain insertion — A de-Pezzer catheter was placed transanally after the creation of the anastomosis, secured to the buttocks, and connected to a urine bag to allow monitoring the amount and the color of the drainage. The catheter was removed on the 3rd day postoperative if the volume collected was insignificant.
  Arms: TD

SUMMARY:
Anastomotic leakage (AL) is considered the commonest major complication after surgery for rectal cancer. Transanal tube drainage role in the prevention of AL is still debatable.

DETAILED DESCRIPTION:
Patients who underwent low or ultralow anterior resection for rectal cancer were enrolled between 01/2015 and 06/2017. A de-Pezzer catheter was placed transanally after the creation of the anastomosis, secured to the buttocks, and connected to a urine bag to allow monitoring the amount and the color of the drainage. The catheter was removed on the 3rd day postoperative if the volume collected was insignificant.

Patients were followed-up on the ward and then in the outpatient's department at two weeks, and one month postoperative. Patients who were suspected to have AL underwent CT with rectal contrast to assess the integrity of the anastomosis. The primary outcome was the incidence of AL. We adopted the definition published by the International Study Group of Rectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Low or ultralow anterior resection with primary anastomosis for biopsy-proven primary rectal cancer

Exclusion Criteria:

* No anastomosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage | 30 days
  Prevention

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Tor Vergata Hospital, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided